CLINICAL TRIAL: NCT00901251
Title: Reproducibility Study of OABSS and Its Response to Treatment - Part 1: Reproducibility -
Brief Title: Reproducibility Study of Over Active Bladder Symptom Score [OABSS]
Acronym: RESORT
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma China, Inc. (Industry)
Responsible Party: Disclosure Director, Astellas Pharma, Inc
Other Study IDs: VESOABCN02
Record Dates: First submitted 2009-05-11; First posted 2009-05-13 (Estimated); Last update posted 2011-03-15 (Estimated); Status verified 2011-03

CONDITIONS: Overactive Bladder
Keywords: OABSS
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
The purpose of this study is to evaluate the reproducibility of over active bladder symptom score (OABSS) in Asian countries.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms OAB for 3 months or longer
* At least 1 urgency episode in last 3 days
* Symptoms of OAB as verified by the screening 3-day bladder diary, defined by:

  * Number of micturition ≥8 times/day
  * Number of urgency episode in 3 days ≥1

Exclusion Criteria:

* Indwelling catheters or practicing intermittent self-catheterization
* Symptomatic urinary tract infection, chronic inflammation
* Diabetic neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Symptomatic OAB patients having urgency episodes
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
OABSS | Weeks of 0 and 2

SECONDARY OUTCOMES:
3-day micturition diary | 2 times in 2-week interval

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma China, Inc.
Locations (5):
- China (5):
  - Beijing
  - Chongqing
  - Shanghai
  - Shenyang
  - Wuhan